CLINICAL TRIAL: NCT04911907
Title: Open, Two-stage, Multicenter, Monotherapy, Phase II Clinical Study of Utidelone Injection in Patients With Advanced or Metastatic Solid Tumors After Failure or Intolerability to Standard Treatment
Brief Title: Clinical Study of Utidelone Injection in Patients With Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Chengdu Biostar Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG01-2002
Record Dates: First submitted 2021-05-30; First posted 2021-06-03 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Squamous cell carcinoma of head and neck: Utidelone Injection (Experimental): Cohort 1 Squamous cell carcinoma of head and neck. Participants will be treated with utidelone monotherapy
  Interventions: Drug: utidelone injection
- Esophageal cancer: Utidelone injection (Experimental): Cohort 2 Esophageal cancer. Participants will be treated with utidelone monotherapy.
  Interventions: Drug: utidelone injection
- Stomach cancer: Utidelone injection (Experimental): Cohort 3 Stomach cancer. Participants will be treated with utidelone monotherapy.
  Interventions: Drug: utidelone injection
- Pancreatic cancer: Utidelone Injection (Experimental): Cohort4 Pancreatic cancer. Participants will be treated with Utidelone monotherapy.
  Interventions: Drug: utidelone injection
- Ovarian cancer: Utidelone Injection (Experimental): Cohort5 Ovarian cancer. Participants will be treated with Utidelone monotherapy.
  Interventions: Drug: utidelone injection
- Cholangiocarcinoma: Utidelone (Experimental): Cohort 6 Cholangiocarcinoma. Participants will be treated with Utidelone monotherapy
  Interventions: Drug: utidelone injection
- Other solid tumors: Utidelone Injection (Experimental): Cohort 7 Other solid tumors. Participants will be treated with Utidelone monotherapy
  Interventions: Drug: utidelone injection

INTERVENTIONS:
Drug: utidelone injection — Utidelone monotherapy 35 mg/m2/day IV transfusing over 90 min. on day 1-day 5 of each 21 day cycle

SUMMARY:
This trial is an open, two-stage, multi-center, phase II clinical trial to evaluate the efficacy and safety of Utidelone in advanced solid tumors (excluding breast cancer, lung cancer, and colorectal cancer) that have failed standard of treatment or were unable to perform standard treatment.

This trial is divided into 2 stages, screening stage and expansion stage. In the screening stage, 10 patients were enrolled for each tumor type(including Squamous cell carcinoma of head and neck, Esophageal cancer, Stomach cancer, Pancreatic cancer, Cholangiocarcinoma, Ovarian cancer and Other solid tumors). Based on the results of the tumor type screening stage, the sponsor and the main investigator will have a discussion and have the alignment of tumor types to enter the expansion stage. The expansion stage will refine the inclusion / exclusion criteria and may adjust the treatment plan based on the tumor type and the combination drug selection. A total of 30-50 patients (including patients enrolled in the screening stage) were enrolled in each specified tumor type during the expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented locally-advanced and/or metastatic solid malignancy (including Squamous cell carcinoma of head and neck, Esophageal cancer, Stomach cancer, Pancreatic cancer, Cholangiocarcinoma, Ovarian cancer and Other solid tumors) that is incurable, and has failed prior standard therapy or for which standard therapy is not appropriate.
2. Have measurable disease based on Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
3. Age 18 -70 years old
4. ECOG performance status of 0-1
5. Life expectancy≥ 3 months
6. Basically normal results from routine blood test within 1 week prior to enrollment

   1. Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
   2. Hemoglobin >= 9 g/dL
   3. Platelets >= 80 x 10^9/L
7. Basically normal liver and renal functions within 1 week prior to enrollment

   1. total bilirubin =< 1.5 x ULN with direct bilirubin within normal range
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (ALT and AST =< 5 x ULN is acceptable if liver metastases are present)
   3. Creatinine clearance>=50 ml/min
8. Women and men of childbearing potential must agree to take effective contraceptive measures during the study and within six months after the last treatment. Female patients must have negative urinary pregnancy test within 7 days before the first treatment (postmenopausal women must have no menstruation for at least 12 months before they are considered unable to conceive)
9. Patients who give written informed consent with good compliance.

Exclusion Criteria:

1. Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks prior to enrollment while participating in this trial, except for the following items:

   1. Nitrosourea or mitomycin C is within 6 weeks before the first dosage of the study drug;
   2. Oral fluorouracil and small molecule targeted drugs are 2 weeks before the first use of the study drug or 5 half-life periods of the drug (whichever is longer);
   3. The traditional Chinese medicine with anti-tumor indication is within 2 weeks before the first use of the research medicine.
2. Received other unlaunched clinical research drugs or treatment within 4 weeks before the first dosage of the research drug.
3. Have undergone major organ surgery (excluding needle biopsy) or experienced significant trauma within 4 weeks prior to the first dosage of study drug, or require elective surgery during the trial period.
4. Symptomatic peripheral neuropathy CTCAE 5.0 grade evaluation ≥ grade 2
5. With severe allergies to castor oil, or have had serious adverse reactions with anti-microtubule drugs in the past
6. Patients of pregnancy or breast feeding
7. Patients with AEs caused by any previous treatment (including systemic and local treatment) that have not yet restored to GRADE 1 (excluding hair loss)
8. Patient with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
9. Patients with active infections and currently need systemic anti-infective treatment
10. Patient with immunodeficiency, including a positive HIV antibody test.
11. Patients with history of active hepatitis B (hepatitis B virus titer> ULN), allow prophylactic antiviral treatment other than interferon; have a history of hepatitis C virus infection (hepatitis C antibody positive).
12. Patients with history of serious cardiovascular and cerebrovascular diseases.
13. Patients with mental disorders or patients with poor compliance.
14. Patients not fitted for this study determined by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Tumor response to utidelone treatment | 12 months from first study treatment
  Reflected by percentage of tumor size reduction or regression, assessed by imaging techniques and expressed as Objective Response Rate (ORR) ORR is defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) according to RECIST. 1.1.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | 12 months from first study treatment
Progression free survival (PFS) | 18 months from first study treatment
  PFS is defined as the duration of time from first study treatment to disease progression or death from any cause as documented by the investigator
Safety profile associated with utidelone injection | 18 months from first study treatment
  Observe and record incidence of Treatment-Emergent Adverse Events and severe adverse effects associated with utidelone injection

CONTACTS AND LOCATIONS:
Overall Officials: JIN LI, MD, Principal Investigator — Shanghai Tongji University Affiliated Oriental Hospital
Locations (3):
- China (3):
  - Luhe Hospital, Capital Medical University, Beijing
  - Obstetrics and Gynecology Hospital, Capital Medical University, Beijing
  - Shanghai East Hospital of Tongji University, Shanghai